CLINICAL TRIAL: NCT01714024
Title: A Molecular and Cellular Comparison of Bone Inductive Properties Of Trabecular Metal® Vs. Titanium Among Healthy, Diabetic, and Osteopenic Subjects
Brief Title: Dental Implant Study Comparing Two Types of Metals Used for Dental Implants
Acronym: ZMU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Zimmer Dental (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: ZMU 11-2539
Record Dates: First submitted 2012-10-17; First posted 2012-10-25 (Estimated); Results first posted 2017-07-12 (Actual); Last update posted 2017-10-12 (Actual); Status verified 2016-01

CONDITIONS: Tooth Replacement
Keywords: Dental; Implant; UNC Dental School; Trabecular Metal; Titanium; Healthy Volunteers; Diabetic; Osteopenic; Bone Inductive Properties; Osseous Healing; GO Health; Offenbacher; Zimmer Dental, Inc.

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Healthy Volunteers (Experimental): Subjects who are non-diabetic, with no history of smoking within the past two years and no metabolic bone disease diagnosis.
  Interventions: Device: Zimmer Trabecular Metal Test Cylinder; Device: Zimmer Titanium Test Cylinder
- Diabetic Subjects (Experimental): Subjects must have Type 2 diabetes mellitus as diagnosed by a physician or in medication history. The condition must be currently diagnosed and treated by medications and/or insulin.
  Interventions: Device: Zimmer Trabecular Metal Test Cylinder; Device: Zimmer Titanium Test Cylinder
- Osteopenic Subjects (Experimental): Subjects must be diagnosed with osteoporosis or osteopenia and must be currently under the care of a physician and treatment with oral bisphosphonates
  Interventions: Device: Zimmer Trabecular Metal Test Cylinder; Device: Zimmer Titanium Test Cylinder

INTERVENTIONS:
Device: Zimmer Trabecular Metal Test Cylinder — For all subjects 2 titanium and 2 trabecular 2.9-3.0 mm x 5 mm test cylinders will be implanted in alveolar bone. One of each type will be removed at 2 weeks. The remaining two will be removed at 4 weeks.
Device: Zimmer Titanium Test Cylinder — For all subjects 2 titanium and 2 trabecular 2.9-3.0 mm x 5 mm test cylinders will be implanted in alveolar bone. One of each type will be removed at 2 weeks. The remaining two will be removed at 4 weeks.

SUMMARY:
The purpose of this research study is to compare the healing differences of two metals (trabecular vs. standard titanium) that are used for dental implants. In addition; investigators will be examine these differences in the gene expression profiles in subjects with three conditions associated with delayed healing: diabetes and osteoporosis.

The study will last at least 11 weeks consisting of 6 appointments. All visits will be carried out at the GO Health Center within the UNC School of Dentistry. Visits will last between 30 minutes to 3 hours depending on the particular visit.

The visits will consist of: Obtaining consent, doing a health history, measuring vital signs, doing dental exams of the teeth and gums, collecting samples of saliva dental radiographs (X-rays), a teeth cleaning, having 4 temporary mini test cylinders placed in areas of the lower jaw where teeth are missing and implant surgery to place up to four permanent implants.

DETAILED DESCRIPTION:
The plan is to recruit subjects into 3 groups: 1) systemically healthy, 2) subjects with diabetes (ADA classification determined by glycosylated hemoglobin A1C levels), and 3) subjects with osteoporosis (limited to those on either no drugs or oral bisphosphonates only). All subjects recruited will have already been approved and treatment planned for implant placement by non-study personnel to avoid any potential conflict of interest. All subjects will have mandibular radiographs that show edentulous ridge areas that provide enough alveolar ridge space to place two test cylinders (each approximately 2.9-3 x 5mm) on each side of the mandible. One side will have two titanium test cylinders and the contralateral side will have two trabecular metal test cylinders. After placement of these 4 test cylinders, one will be removed contra laterally from each side at weeks 2 and 4 of healing. Thus, by 28 days all test cylinders will be removed.

It has been our experience that each cylinder after removal will contain enough cells to provide approximately 10-20μg of total RNA. This quantity of total RNA is sufficient to run an Affymetrix chip and have enough mRNA for PCR confirmation. Sampling at 3 days after placement is too soon, as it does not provide adequate mRNA for the analysis, since the clot has not become remodeled or adequately organized to be cellular. Thus, by 1 week organization of the osseous healing will have begun and at week 2 it will be beginning to mature. The week 2 sampling time point) will provide us with early molecular kinetics of the healing response to compare the two metal surfaces and the differences in gene expression that may be associated with diabetes and osteoporosis. At weeks 2 and 4 the test cylinders will be removed using a 5.0 mm diameter tissue punch and a 5 mm trephine drill. Investigators will select 18 random patients (6 subjects per group) to provide (two test cylinders for each, 36 samples) for histology. Investigators will use the trephine drill to remove the 4 week test cylinders in all 3 groups of subjects. In all cases, a subject is eligible for this study by being pretreatment planned to receive a permanent implant bilaterally, which will be placed at donor sites. According to the participant's individual treatment plan, after test cylinders are removed, each site will receive an implant using either a standard 4.1 or 4.7 mm tapered screw vent design implant. The removed test cylinders will be briefly rinsed in saline and prepared chair side for either mRNA extraction or for histology.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be adult males or females age 21 to 80 years (inclusive).
* Subjects must be able and willing to follow study procedures and instructions in English.
* Subjects must have read, understood and signed an informed consent form in English.
* Subjects must have at least four mandibular implants as their future treatment needs.

Subjects must meet one of the following categories to be considered for enrollment:

* Group 1 (control): Subjects must be non-diabetic, no history of smoking within the last two years and no metabolic bone disease diagnosis.
* Group 2 (diabetic): Subjects must have Type 2 diabetes mellitus as diagnosed by a physician or in medication history. The condition must be currently diagnosed and treated by medications and/or insulin. An HbA1C test performed either within past 3 months must be available or one will be done at the first visit by study personnel. Subjects must have no history of smoking within the last two years nor have any diagnosis of metabolic bone disease.
* Group 3 (Osteoporosis or osteopenia): Subjects must be diagnosed with osteoporosis or osteopenia and must be currently under the care of a physician and treatment with oral bisphosphonates. Subjects must have never had intravenous (IV) bisphosphonates. Subjects in this group must be non-diabetic and no history of smoking within the last 2 years.

Subjects undergoing test cylinder placement should be in adequate periodontal health prior to implant placement. This includes having probing depth ≤ 4 mm for all remaining teeth at the same quadrant of the proposed cylinder placement. Patients with periodontal probing sites with probing depths of up to 5 mm may also be included if bleeding on probing in these sites is absent. Each subject should be considered to be periodontally stable prior to receiving test cylinders.

Exclusion Criteria:

* Individuals who have a chronic disease with oral manifestations.
* Individuals who exhibit gross oral pathology.
* The use of either antibiotics or chronic use of NSAIDs within 1 month prior to screening examination.
* Individuals that require antibiotic prophylaxis prior to dental treatment.
* Chronic treatment (i.e. two weeks or more) with any medication known to affect periodontal status (e.g. phenytoin, calcium antagonists, cyclosporine, Coumadin) within 1 month prior to screening examination.
* Systemic conditions, except diabetes, osteoporosis and osteopenia that are known to affect periodontal status.
* Individual with uncontrolled parafunctional habits, such as clenching and bruxing on objects, that could adversely impact implant survival
* Individuals with a history of intravenous bisphosphonates Individuals with active infectious diseases such as hepatitis, HIV or tuberculosis.
* Individuals with a current tobacco use history.
* Individuals who are known to be pregnant, breastfeeding or planning to become pregnant within 3 months.
* Individuals with blood disorders and /or currently taking anticoagulants medications, unless he or she can provide a current International normalized ratio (INR) showing normal (0.8 - 2.0) values.
* Individuals receiving any therapy known to affect healing, such as high dose corticosteroids, radiation therapy or chemotherapy.
* Individuals allergic to topical or local anesthesia

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2012-10; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Offenbacher, DDS, PhD, MMSc, Principal Investigator — University of North Carolina School of Dentistry
Locations (1):
- General & Oral Health Center, Chapel Hill, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Healthy Volunteers | Diabetic Subjects | Osteopenic Subjects
Started | 13 | 18 | 11
Completed | 12 | 12 | 8
Not Completed | 1 | 6 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Volunteers | Diabetic Subjects | Osteopenic Subjects | Total
Number analyzed (Participants) | 12 | 12 | 8 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 5 | 3 | 16
  >=65 years | 4 | 7 | 5 | 16
Age, Continuous [Mean (Full Range); unit: years] | 59.33 [39 to 75] | 64.33 [54 to 71] | 66.38 [59 to 76] | 64.22 [39 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 8 | 20
  Male | 5 | 7 | 0 | 12
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 12 | 36

OUTCOME MEASURES:

1. Primary Outcome: Fold Change in Gene Expression Comparing Trabecular Metal to Standard Titanium.
Description: Samples were analyzed comparing the osteogenic potential associated with titanium and porous tantalum dental implants (cylinders) at 2 and 4 weeks using transcriptome analyses. The primary outcome data are displayed showing the Average Delta ∆ (Ct) for osteogenic genes relative to the housekeeping markers. The numerical value of the CT is inversely related to the amount of amplicon in the reaction (i.e., the lower the CT, the greater the amount of amplicon).
Time Frame: 2 weeks & 4 weeks post placement
Measure: Mean (Standard Deviation); unit: Average Delta ∆ (Ct)
Groups:
- Healthy/Tantalum; Healthy/Titanium: Subjects who are non-diabetic, with no history of smoking within the past two years and no metabolic bone disease diagnosis.
  For all subjects 2 titanium and 2 trabecular 2.9-3.0 mm x 5 mm test cylinders were implanted in alveolar bone. One of each type will be removed at 2 weeks. The remaining two were removed at 4 weeks.
- Osteopenic/Tantalum; Osteopenic/Titanium: Subjects must be diagnosed with osteoporosis or osteopenia, non-diabetic, with no history of smoking within the past two years
  For all subjects 2 titanium and 2 trabecular 2.9-3.0 mm x 5 mm test cylinders were implanted in alveolar bone. One of each type will be removed at 2 weeks. The remaining two were removed at 4 weeks.
- Diabetic/Tantalum; Diabetic/Titanium: Subjects who are diabetic, with no history of smoking within the past two years and no metabolic bone disease diagnosis
  For all subjects 2 titanium and 2 trabecular 2.9-3.0 mm x 5 mm test cylinders were implanted in alveolar bone. One of each type will be removed at 2 weeks. The remaining two were removed at 4 weeks.
Arm/Group | Healthy/Tantalum | Healthy/Titanium | Osteopenic/Tantalum | Osteopenic/Titanium | Diabetic/Tantalum | Diabetic/Titanium
Number analyzed (Participants) | 12 | 12 | 8 | 8 | 12 | 12
Average Delta ∆ (Ct)
  BMP2 (2 weeks) | 7.6758 (0.12) | 9.2208 (1.15) | 4.6085 (2.67) | 5.2331 (1.69) | 7.1463 (1.67) | 6.5207 (1.73)
  DLX5 (2 week) | 10.4258 (.038) | 12.2275 (1.08) | 5.9966 (1.56) | 6.1543 (1.75) | 9.4077 (1.09) | 9.4038 (1.12)
  BMP1 (2 weeks) | 4.2225 (0.46) | 5.9042 (0.84) | 1.8624 (1.49) | 2.4895 (1.31) | 3.9986 (1.77) | 3.5056 (1.57)
  BGN (2 Weeks) | 0.6525 (0.63) | 3.0942 (1.25) | -1.9201 (0.31) | -0.6761 (0.22) | 0.9032 (1.86) | .03906 (2.30)
  COL14A1 (2 weeks) | 2.9192 (0.52) | 4.4442 (0.33) | 0.5529 (0.42) | 0.9162 (0.66) | 2.4111 (1.31) | 3.0112 (1.18)
  CSF1 (2 weeks) | 5.2292 (0.51) | 6.4042 (0.23) | 0.8180 (0.95) | 2.1533 (0.81) | 4.5506 (1.39) | 4.6397 (1.21)
  GLI1 (4 weeks) | 5.7365 (0.27) | 8.2807 (0.23) | 4.8091 (0.33) | 4.7381 (1.41) | 8.7988 (3.77) | 9.1999 (2.04)
  IGF1R (4 weeks) | 1.5259 (0.31) | 3.8134 (1.08) | 2.6811 (1.08) | 3.0398 (0.30) | 5.6048 (2.31) | 6.3467 (0.65)
  PHEX (4 weeks) | 2.1578 (0.58) | 6.4186 (2.08) | 0.2916 (0.26) | 3.9890 (0.41) | 5.7960 (1.62) | 6.8678 (0.80)
  FGF1 (4 weeks) | 4.0907 (0.19) | 5.3543 (0.85) | 2.5977 (0.23) | 3.1967 (1.77) | 6.3124 (4.51) | 5.8513 (0.53)
  FGFR2 (4 weeks) | 1.5910 (0.38) | 3.8245 (1.98) | 0.8745 (0.10) | 2.9709 (0.34) | 4.3674 (2.19) | 5.4090 (0.71)
  TGFBR2 (4weeks) | 0.3029 (0.25) | 0.9102 (0.79) | -0.9658 (1.74) | -0.2509 (2.96) | 2.2868 (1.89) | 2.9935 (1.23)
  FGF2 (4 weeks) | 4.7981 (0.26) | 5.9102 (0.71) | -0.9658 (1.33) | 4.2644 (1.97) | 6.8459 (3.20) | 7.7363 (1.34)
  FGFR1 (4 weeks) | 0.3229 (0.71) | 1.4584 (0.41) | -0.5135 (0.20) | -0.9003 (0.24) | 2.4234 (2.36) | 2.7818 (2.16)
  IGF1 (4 weeks) | 0.5603 (1.09) | 3.3670 (1.25) | 2.1275 (2.47) | 1.8615 (0.40) | 4.2738 (1.55) | 5.4869 (1.68)
  BMP2 (4 weeks) | 7.0738 (1.26) | 4.3821 (0.50) | 3.3444 (1.30) | 3.6476 (0.94) | 7.1463 (2.56) | 6.5207 (0.91)
  BMP1 (4 weeks) | 3.6543 (0.43) | 2.2410 (0.59) | 0.6949 (0.14) | 1.0592 (0.20) | 3.9986 (2.71) | 1.5697 (1.63)

2. Secondary Outcome: Group Based Differences (i.e. Healthy, Osteopenic and Diabetic) in Gene Expression Using Fold Changes Between Titanium and Trabecular at 4 Weeks.
Description: Findings from expression arrays will be used to perform quantitative PCR analyses using SAB Superarrays (SuperArray GEArray), to enable a quantitativeassay of mRNA levels of specific inflammatory and growth factor molecules
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: Fold Change
Groups:
- Healthy Tantalum; Heathy Titanium: Subjects who are non-diabetic, with no history of smoking within the past two years and no metabolic bone disease diagnosis.
  Zimmer Metal Test Cylinder: For all subjects 2 titanium and 2 trabecular 2.9-3.0 mm x 5 mm test cylinders will be implanted in alveolar bone. One of each type will be removed at 2 weeks. The remaining two will be removed at 4 weeks.
- Diabetic Tantalum; Diabetic Titanium: Subjects must have Type 2 diabetes mellitus as diagnosed by a physician or in medication history. The condition must be currently diagnosed and treated by medications and/or insulin.
  Zimmer Metal Test Cylinder: For all subjects 2 titanium and 2 trabecular 2.9-3.0 mm x 5 mm test cylinders will be implanted in alveolar bone. One of each type will be removed at 2 weeks. The remaining two will be removed at 4 weeks
- Osteoporosis Tantalum; Osteoporosis Titanium: Subjects must be diagnosed with osteoporosis or osteopenia and must be currently under the care of a physician and treatment with oral bisphosphonates
  Zimmer Metal Test Cylinder: For all subjects 2 titanium and 2 trabecular 2.9-3.0 mm x 5 mm test cylinders will be implanted in alveolar bone. One of each type will be removed at 2 weeks. The remaining two will be removed at 4 weeks.
Arm/Group | Healthy Tantalum | Heathy Titanium | Diabetic Tantalum | Diabetic Titanium | Osteoporosis Tantalum | Osteoporosis Titanium
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 8 | 8
Fold Change
  PHEX | 2.158 (0.58) | 6.419 (2.08) | 5.796 (1.62) | 6.868 (0.80) | 0.292 (0.26) | 3.989 (0.41)
  FGF1 | 40.91 (0.19) | 5.3454 (0.85) | 6.312 (4.51) | 5.851 (0.53) | 2.598 (0.23) | 3.197 (1.77)
  FGFR2 | 1.591 (0.38) | 3.824 (1.98) | 4.367 (2019) | 5.409 (0.71) | 0.875 (0.10) | 2.971 (0.34)
  TGFBR2 | 0.303 (0.25) | 0.901 (0.79) | 2.287 (1.89) | 2.994 (1.23) | -0.966 (1.74) | -0.251 (2.96)
  FGF2 | 4.79 (0.26) | 5.910 (0.71) | 6.846 (3.20) | 7.736 (1.34) | -0.966 (1.33) | 4.264 (1.97)
  FGFR1 | 0.323 (0.71) | 1.458 (0.41) | 2.423 (2.36) | 2.782 (2.16) | -0.513 (0.20) | -0.9 (0.24)
  IGF1 | 0.56 (1.09) | 3.367 (1.25) | 4.2474 (1.55) | 5.487 (1.68) | 2.128 (2.47) | 1.861 (0.4)
  BMP2 | 7.074 (1.26) | 4.382 (0.5) | 7.146 (2.56) | 6.521 (0.91) | 3.344 (1.30) | 3.648 (0.94)
  BMP1 | 3.654 (0.43) | 2.241 (0.59) | 3.999 (2.71) | 1.570 (1.63) | 0.695 (0.14) | 1.059 (0.2)
  CSF1 | 5.229 (0.51) | 6.404 (0.23) | 4.551 (1.39) | 4.64 (1.21) | 0.818 (0.95) | 2.153 (0.81)
  GLI1 | 5.736 (0.27) | 8.281 (0.23) | 8.799 (3.77) | 9.2 (2.04) | 4.809 (0.33) | 4.738 (1.41)
  IGF1R | 1.526 (0.31) | 3.813 (1.08) | 5.605 (2.31) | 6.347 (0.65) | 2.681 (1.08) | 3.04 (0.30)

ADVERSE EVENTS:
Time Frame: 2 years, 4 months
Arm/Group | Healthy Volunteers | Diabetic Subjects | Osteopenic Subjects
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/8
Other Adverse Events (participants affected / at risk) | 2/12 | 0/12 | 2/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthy Volunteers (N=12) | Diabetic Subjects (N=12) | Osteopenic Subjects (N=8)
Gingival Swelling & Pain (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Delayed healing response (General disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No